CLINICAL TRIAL: NCT01593904
Title: Venous Irregularities, Flow and Perfusion in MS Study
Acronym: VERIFYMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Synergy Health Concepts, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VERIFYMS
Record Dates: First submitted 2012-05-06; First posted 2012-05-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Venous Irregularities, Flow and Perfusion in MS and Non-MS Participants
Keywords: CCSVI, Flow, Perfusion in MS

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
1. What is the true incidence of CCSVI in patients with MS in a study comparing MRI on MS patients and controls.
2. Are the beneficial outcomes from treatment placebo? By measuring changes in brain perfusion and Cerebrospinal flow before and after the procedure on a large number of patients to determine these outcomes

DETAILED DESCRIPTION:
The purpose of this study is to compare a MS subject to a non-MS, non-blood related subject. The 3D structural information provided by the protocol combined with the ability to observe and quantify flow through the major vessels of the neck, as well as the azygous vein, make it an ideal method for evaluating subjects' venous outflow. The protocol also has the potential to confirm the diagnosis of Multiple Sclerosis, observe any changes in the parenchyma, as well as provide data on any potential co-morbidity which may have been previously overlooked or non-emergent. The baseline scan data acquired on normal and pre-treatment MS patients can be tracked longitudinally for MSpatients for changes in: arterial and venous cross sectional area; morphological changes of vessels, brain structures, and lesions; flow distribution and flow patterns in arteries, veins, and cerebrospinal fluid (CSF); iron quantification in the deep basal ganglia and thalamus; parenchymal lesion volume and morphology; atrophy or ratio of gray matter, white matter; and CSF in the intracranial space; and appearance of intracranial veins and potential iron lesions in the parenchyma. A major benefit is that MRI is independent of operator bias and acquisition can be easily reproduced.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend the nature of the study, including the risks and benefits
* Ability to execute an informed consent
* Males or Females between the ages of 20 and 65 years of age
* Voluntary agreement to participate in the study: Venous Irregularities, Flow and Perfusion in MS study (VERIFY MS Study)

Exclusion Criteria:

* Any implantable/metallic objects that prevents subject from having a magnetic resonance imaging (MRI/MRV) study.
* Any person who has a contraindication to contrast administration.
* History of claustrophobia
* Special Populations. Special groups include, but are not limited to children, prisoners, pregnant women, fetuses, and cognitively impaired individuals who are unable to provide informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Human subjects will be approached for participation in this study that are receiving or seeking medical care at Synergy Health Concepts Inc.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-01; Study Completion 2013-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John Joseph Hewett, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Synergy Health Concepts Inc., Newport Beach, California, United States